CLINICAL TRIAL: NCT03495648
Title: Tanglewood Trail Walking Program to Increase Phytonutrient Intake and Physical Activity in a Rural Kentucky Town
Brief Title: Tanglewood Trail Walking Program in Rural Kentucky 2017
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dawn Brewer (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor-Investigator, Dawn Brewer, Assistant Professor, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 17-0283-P2H 2017; P42ES007380 (NIH)
Record Dates: First submitted 2018-03-19; First posted 2018-04-12 (Actual); Results first posted 2021-11-17 (Actual); Last update posted 2021-11-17 (Actual); Status verified 2021-11

CONDITIONS: Dietary Habits
Keywords: farmers market; Appalachia; physical activity; fruit and vegetable voucher program
MeSH Terms: conditions — Feeding Behavior; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Walking Group (Low Engagers) (Experimental): Subjects will participate in a walking group led by a community organizer as a means to get to a local farmer's market. Low engagers are defined as those participants who walked to the market two or fewer times during the program.
  Interventions: Behavioral: walking group led by a community organizer
- Walking Group (High Engagers) (Experimental): Subjects will participate in a walking group led by a community organizer as a means to get to a local farmer's market. High engagers are defined as those participants who walked to the market three or more times during the program.
  Interventions: Behavioral: walking group led by a community organizer

INTERVENTIONS:
Behavioral: walking group led by a community organizer — Subjects will walk 1 kilometer from a pre-determined point to a local farmer's market.

SUMMARY:
The Tanglewood Trail Walking Program is a well-established community health initiative that encourages community members to walk approximately 1 mile to the Whitesburg Farmers Market each Saturday. The study aims to determine if walking to the market with a community health coach results in healthier options being selected at the market.

DETAILED DESCRIPTION:
In the summer of 2017, community members of Whitesburg, KY were recruited to join the Tanglewood Trail Walking Program to the Whitesburg farmers market. Each Saturday, participants reported whether or not they walked the 1-mile trail to the farmers market and they reported which fruits and vegetables they purchased. The Walking Program was held June - Sept 2017. Participants completed questionnaires about fruit and vegetable consumption and physical activity. Participants also provided physical and biological measurements.

Although originally designed to compare data among walkers and non-walkers, the protocol was changed due to participant feasibility. Data were analyzed by comparing "low engagers" - those who walked to the market fewer than three times during the program - or "high engagers" - those who walked three or more times during the program. Data were collected at baseline and 3 months.

The data for years 2019 and 2020 of the Tanglewood to Trail walking program are registered separately in ClinicalTrials.gov.

ELIGIBILITY:
Inclusion Criteria:

* ability to walk 1 kilometer

Exclusion Criteria:

* pregnant
* institutionalized adults
* impaired consent ability
* prisoners

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2020-09-24 (Actual); Study Completion 2020-09-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Brewer, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No
No current plan to share data.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 123 participants were enrolled, but two participants dropped out of the study within the first month due to lack of interest.
Period: Overall Study
Arm/Group | Walking Group (Low Engagers) | Walking Group (High Engagers)
Started | 60 | 61
Completed | 60 | 61
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Walking Group (Low Engagers) | Walking Group (High Engagers) | Total
Number analyzed (Participants) | 60 | 61 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (14.7) | 46.7 (14.7) | 50.2 (15.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 37 | 72
  Male | 25 | 24 | 49
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 58 | 58 | 116
  Unknown or Not Reported | 2 | 3 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 57 | 59 | 116
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 60 | 61 | 121
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.4 (7.3) | 33.4 (7.0) | 33.4 (7.1)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 80.6 (9.3) | 84.3 (10.8) | 82.5 (10.2)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 128.4 (15.7) | 129.1 (18.0) | 128.8 (16.9)
Total Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 168.6 (34.8) | 169.1 (37.4) | 168.8 (36.0)
LDL Cholesterol [Mean (Standard Deviation); unit: mg/dL] | 93.0 (25.9) | 92.4 (27.3) | 92.7 (26.5)
Total Cholesterol/HDL Ratio [Mean (Standard Deviation); unit: ratio] | 4.2 (1.7) | 4.1 (1.5) | 4.1 (1.6)
Hemoglobin A1c [Mean (Standard Deviation); unit: percentage of glycosylated hemoglobin] | 6.2 (1.3) | 6.2 (1.4) | 6.2 (1.4)
ASCVD (Atherosclerotic Cardiovascular Disease) Risk [Mean (Standard Deviation); unit: risk] — The ASCVD (atherosclerotic cardiovascular disease) risk is a national guideline developed by the American College of Cardiology. It is a calculation of the 10-year risk of having a cardiovascular problem, such as a heart attack or stroke. This risk estimate considers age, sex, race, cholesterol levels, blood pressure, medication use, diabetic status, and smoking status, with a range from 0 to >20. Lower scores indicate lower risk of cardiovascular disease.
  risk | 11.2 (14.2) | 9.1 (10.0) | 10.2 (12.4)

OUTCOME MEASURES:

1. Primary Outcome: Change in Carotenoid Levels Over Time
Description: Subjects' carotenoid status will be measured using a carotenoid Raman Spectroscopy to determine if walking combined with a voucher for fruits and vegetables increases intake in fruits and vegetables as measured by carotenoid status.
Time Frame: Baseline and 3 months
Population: No data were collected for this outcome measure.
Arm/Group | Walking Group (Low Engagers) | Walking Group (High Engagers)
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in A1c
Description: Subjects' A1c will be measured to determine if walking combined with a voucher for fruits and vegetables changes participant A1c. Data were collected at baseline and 3 months and the difference will be calculated.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Walking Group (Low Engagers) | Walking Group (High Engagers)
Number analyzed (Participants) | 36 | 51
percent change | -0.31 (0.53) | -0.20 (0.52)

3. Secondary Outcome: Change in LDL Cholesterol
Description: Subjects' LDL will be measured to determine if walking combined with a voucher for fruits and vegetables changes participant LDL.
Time Frame: Baseline and 3 months
Population: Not all participants completed this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Walking Group (Low Engagers) | Walking Group (High Engagers)
Number analyzed (Participants) | 39 | 50
mg/dL | -11.9 (23.8) | -12.7 (17.5)

4. Secondary Outcome: Change in HDL Cholesterol
Description: Subjects' HDL will be measured to determine if walking combined with a voucher for fruits and vegetables changes participant HDL.
Time Frame: Baseline and 3 months
Population: Data are shown by sex: low engagers (10 males and 24 females) and high engagers (11 male and 37 female). Not all participants completed this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Walking Group (Low Engagers) | Walking Group (High Engagers)
Number analyzed (Participants) | 34 | 48
mg/dL
  Males: number analyzed (Participants) | 10 | 11
  Males | 1.6 (4.3) | 8.8 (7.2)
  Females: number analyzed (Participants) | 24 | 37
  Females | 0.04 (8.5) | 5.3 (10.0)

5. Secondary Outcome: Change in Total Cholesterol
Description: Subjects' total cholesterol will be measured to determine if walking combined with a voucher for fruits and vegetables changes participant total cholesterol.
Time Frame: Baseline and 3 months
Population: Not all participants completed this outcome measure.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Walking Group (Low Engagers) | Walking Group (High Engagers)
Number analyzed (Participants) | 39 | 50
mg/dL | -14.8 (32.5) | -11.0 (24.2)

6. Secondary Outcome: Change in Weight
Description: Subjects' weight will be measured to determine if walking combined with a voucher for fruits and vegetables changes participant weight.
Time Frame: Baseline and 3 months
Population: Not all participants completed this outcome measure.
Measure: Mean (Standard Deviation); unit: lb
Arm/Group | Walking Group (Low Engagers) | Walking Group (High Engagers)
Number analyzed (Participants) | 40 | 51
lb | 0.23 (5.4) | -1.4 (11.8)

7. Secondary Outcome: Change in Waist Circumference
Description: Subjects' waist circumference will be measured to determine if walking combined with a voucher for fruits and vegetables changes participant waist circumference.
Time Frame: Baseline and 3 months
Population: Data are shown by sex: low engagers (10 male and 25 female) and high engagers (11 male and 39 female). Not all participants completed this outcome measure.
Measure: Mean (Standard Deviation); unit: inches
Arm/Group | Walking Group (Low Engagers) | Walking Group (High Engagers)
Number analyzed (Participants) | 35 | 50
inches
  Male: number analyzed (Participants) | 10 | 11
  Male | -0.30 (1.3) | -0.34 (2.1)
  Female: number analyzed (Participants) | 25 | 39
  Female | -0.33 (2.3) | -0.88 (3.8)

8. Secondary Outcome: Change in Self-reported Activity Level
Description: Subjects' self-reported activity level will be measured as self-reported days of leisure physical activity per week.
Time Frame: Baseline and 3 months
Population: Not all participants completed this outcome measure.
Measure: Mean (Standard Deviation); unit: days of physical activity per week
Arm/Group | Walking Group (Low Engagers) | Walking Group (High Engagers)
Number analyzed (Participants) | 26 | 35
days of physical activity per week | 1.7 (2.6) | 1.4 (2.1)

9. Secondary Outcome: Change in Self-reported Fruit and Vegetable Intake
Description: Subjects' self-reported total servings of fruit and vegetable intake per day.
Time Frame: Baseline and 3 months
Population: Not all participants completed this outcome measure.
Measure: Mean (Standard Deviation); unit: servings of fruit and vegetables per day
Arm/Group | Walking Group (Low Engagers) | Walking Group (High Engagers)
Number analyzed (Participants) | 25 | 37
servings of fruit and vegetables per day | 1.0 (4.2) | 2.4 (2.7)

10. Secondary Outcome: Group Cohesion
Description: Subjects' group cohesion was measured post-intervention using the Physical Activity Group Environment Questionnaire" (also known as PAGE-Q). There are 20 questions, ranked using a Likert Scale with 1 being "strongly disagree" and 9 "strongly agree." Scores range from 20-180; higher scores indicate more social cohesion.
Time Frame: 3 months
Population: Not all participants completed this outcome measure.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Walking Group (Low Engagers) | Walking Group (High Engagers)
Number analyzed (Participants) | 20 | 36
score on a scale | 130.2 (53.1) | 155.3 (40.7)

11. Secondary Outcome: Understanding of Plant-based Phytonutrients
Description: Participants will be asked a question demonstrating their understanding of the importance of ingesting plant-based nutrients. Possible answers are yes, no, or not sure. Data will be presented as the number of participants in each group that understood the importance of plant-based nutrients.
Time Frame: 3 months
Population: Not all participants completed the questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Walking Group (Low Engagers) | Walking Group (High Engagers)
Number analyzed (Participants) | 52 | 55
Participants
  baseline | 11 | 17
  3 months: number analyzed (Participants) | 24 | 35
  3 months | 12 | 20

12. Secondary Outcome: Belief in the Benefit of Plant-based Nutrients
Description: Participants will be asked a question demonstrating their appreciation of plant-based nutrients. Possible answers are yes, no, or not sure. Data will be presented as the number of participants in each group that understood the importance of plant-based nutrients.
Time Frame: 3 months
Population: Not all participants completed the questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Walking Group (Low Engagers) | Walking Group (High Engagers)
Number analyzed (Participants) | 25 | 28
Participants
  baseline | 7 | 12
  3 months: number analyzed (Participants) | 16 | 24
  3 months | 5 | 19

13. Secondary Outcome: Belief in the Preventative Effects of Plant-Based Nutrients
Description: Participants will be asked a question demonstrating their beliefs of plant-based nutrients. Possible answers are yes, no, or not sure. Data will be presented as the number of participants in each group that understood the importance of plant-based nutrients.
Time Frame: 3 months
Population: Not all participants completed the questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Walking Group (Low Engagers) | Walking Group (High Engagers)
Number analyzed (Participants) | 24 | 27
Participants
  baseline | 8 | 11
  3 months: number analyzed (Participants) | 14 | 23
  3 months | 11 | 18

14. Secondary Outcome: Belief in the Role of Healthy Diet in Protecting Health From Pollutants
Description: Participants will be asked a question demonstrating their beliefs that a healthy diet might protect health from environmental pollutants. Possible answers are yes, no, or not sure. Data will be presented as the number of participants in each group that understood the importance of a healthy diet.
Time Frame: 3 months
Population: Not all participants completed the questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Walking Group (Low Engagers) | Walking Group (High Engagers)
Number analyzed (Participants) | 23 | 27
Participants
  baseline | 6 | 9
  3 months: number analyzed (Participants) | 15 | 24
  3 months | 9 | 15

15. Secondary Outcome: Knowledge of Which Foods Contain Phytonutrients
Description: Participants will be asked a question about which foods contain phytonutrients. Possible answers are meat, dairy, plant foods, all foods, or don't know. Data will be presented as the number of participants in each group that correctly identified plant foods.
Time Frame: 3 months
Population: Not all participants completed the questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Walking Group (Low Engagers) | Walking Group (High Engagers)
Number analyzed (Participants) | 56 | 56
Participants
  baseline | 17 | 17
  3 months: number analyzed (Participants) | 25 | 35
  3 months | 13 | 27

16. Secondary Outcome: Knowledge of Environmental Pollutants
Description: Participants will be asked to identify environmental pollutants from a list. Possible answers are polychlorinated biphenyls (PCBs), mercury, nitrites, all of those, none of those, or don't know. Data will be presented as the number of participants in each group that correctly identified all of those.
Time Frame: 3 months
Population: Not all participants completed the questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Walking Group (Low Engagers) | Walking Group (High Engagers)
Number analyzed (Participants) | 49 | 51
Participants
  baseline | 13 | 22
  3 months: number analyzed (Participants) | 24 | 36
  3 months | 8 | 15

ADVERSE EVENTS:
Time Frame: Adverse event data were not collected during the course of this study.
Description: Adverse event and mortality data were not collected during the course of this study.
Arm/Group | Walking Group (Low Engagers) | Walking Group (High Engagers)
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2017-05-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT03495648/Prot_SAP_ICF_000.pdf